CLINICAL TRIAL: NCT01542541
Title: A Clinical Study to Limit Physiologic Intestinal FDG Uptake Uptake on PET-CT Scans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Alan C. Moss, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010P000101
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Intestinal FDG Uptake
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin (Experimental)
  Interventions: Drug: Rifaximin
- Control (No Intervention): Randomly-selected matched PET-CT scans performed on same day as intervention group.

INTERVENTIONS:
Drug: Rifaximin — 550mg BID for 2 days
  Other Names: Xifaxan
  Arms: Rifaximin

SUMMARY:
Patients who undergo PET-CT scans to look for cancer are given an intravenous contrast (FDG) that is taken-up by active cells such as cancer cells. This contrast can then be seen in the body using the PET-CT scanner. However, cells in the colon also take up the FDG, and can produce "false positive" signals from the colon. Our hypothesis is that much of this signal comes from bacteria that are present in high concentrations in the colon. If this is the case, using an antibiotic to suppress the activity of bacteria may improve the ability of PET-CT to distinguish abnormal cells from normal cells in the colon.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically-indicated PET-CT scan for non-GI lymphoma

Exclusion Criteria:

* Patients with known Inflammatory Bowel Disease
* Patients with known colon cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifaximin | Control
Started | 38 | 30
Completed | 30 | 30
Not Completed | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifaximin | Control | Total
Number analyzed (Participants) | 38 | 30 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (19) | 56 (19) | 56 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 21 | 15 | 36
Region of Enrollment [Number; unit: participants]
  United States | 38 | 30 | 68

OUTCOME MEASURES:

1. Primary Outcome: SUVmax of FDG in Each Colonic Segment
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Rifaximin | Control
Number analyzed (Participants) | 30 | 30
SUV | 4.6 (2.3) | 4.3 (2.7)

2. Secondary Outcome: SUVavg in Each Colonic Segment
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Rifaximin | Control
Number analyzed (Participants) | 30 | 30
SUV | 1.6 (0.9) | 1.8 (0.9)

ADVERSE EVENTS:
Arm/Group | Rifaximin | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less